CLINICAL TRIAL: NCT01006928
Title: Association Between the Support of Neonatal Intensive Care Unit (NICU) Team and Subjective Health of Parents to a Premature Infant
Brief Title: Association Between the Support of NICU Team and Subjective Health of Parents
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Erez Nadir, MD, Hillel Yaffe medical center
Other Study IDs: HY0015-09-IL
Record Dates: First submitted 2009-11-01; First posted 2009-11-03 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Conditions Influencing Health Status
Keywords: Subjective health feeling; NICU; team support

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mothers: Mother of infants in NICU
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — Questionaire to mothers

SUMMARY:
Preterm birth is a traumatic event for parents. They cope with threatening and unfamiliar environment of hospital, losing the parental role, and frustration. The NICU team is the main support source for these parents. Support and providing information are most important for parents, as they can have some control, involvement and self confidence during the hospitalization, and also feel healthier. The hypothesis of this study is that better support to parents lead to better subjective health feeling by them.

The study will be held among mothers to infants in NICU who are at least 7 days old. The study will use a questionaire to assess the subjective health feeling and the estimation of the support from the team. Sample size is about 150 mothers.

DETAILED DESCRIPTION:
Preterm birth is a traumatic event for parents. They cope with threatening and unfamiliar environment of hospital, losing the parental role, and frustration. The NICU team is the main support source for these parents. Support and providing information are most important for parents, as they can have some control, involvement and self confidence during the hospitalization, and also feel healthier. The hypothesis of this study is that better support to parents lead to better subjective health feeling by them.

The study will be held among mothers to infants in NICU who are at least 7 days old. The study will use a questionaire to assess the subjective health feeling and the estimation of the support from the team. Sample size is about 150 mothers.

ELIGIBILITY:
Inclusion Criteria:

* Mothers to preterm infants in NICU

Exclusion Criteria:

* Mothers to Infants in NICU who are not preterm
* Mothers to Infants in NICU who died during hospitalization
* Mothers to Infants in NICU who were transferred to another hospital during hospitalization

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Mothers of infants in NICU
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Good subjective health feeling of mother. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe medical centet, Hadera, Israel
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel, Israel

REFERENCES:
- [Background] Arockiasamy V, Holsti L, Albersheim S. Fathers' experiences in the neonatal intensive care unit: a search for control. Pediatrics. 2008 Feb;121(2):e215-22. doi: 10.1542/peds.2007-1005. Epub 2008 Jan 8. PMID 18182470
- [Background] Bloom KC. The development of attachment behaviors in pregnant adolescents. Nurs Res. 1995 Sep-Oct;44(5):284-9. PMID 7567484